CLINICAL TRIAL: NCT04111393
Title: Transoral Removal of Specimen During Laparoscopic Gastric Resection
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, cihan gokler, Inonu, Inonu University
Other Study IDs: 2019/2-4
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2014-01

CONDITIONS: Gastric Disease; Bariatric Surgery Candidate
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: transoral specimen extraction — transoral specimen extraction during laparoscopic gastric resection
  Other Names: laparoscopic gastric resection

SUMMARY:
Investigators aimed to present the patients who underwent laparoscopic gastrectomy with transoral specimen extraction.

DETAILED DESCRIPTION:
Minimally invasive surgical procedures such as NOSE (Natural orifice spesmen extraction) and NOTES (Natural orifice translumenal endoscopic surgery) are gradually increasing. The transoral way is probably the least used for NOSE.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic gastric resection
* Patients aged 18-70 years

Exclusion Criteria:

* other transorally removed organs (appendix, gallbladder, surrenal)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent sleeve gastrectomy for morbid obesity, subtotal gastrectomy for pyloric obstruction, and extensive gastric resection for gastrointestinal stromac tumor
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-28 (Actual)

PRIMARY OUTCOMES:
Transoral Specimen Extraction During Laparoscopic Gastric Resection | 2 years
  laparoscopic gastric resections due to sleeve gastrectomy or pyloric obstruction will be observed after transoral removal.

CONTACTS AND LOCATIONS:
Locations (1):
- Cihan Gokler, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The patients who underwent laparoscopic gastric resection with transoral extraction between 2014-2018 in Inonu University gastroenterology surgery clinic will be evaluated retrospectively. Patients will be evaluated in terms of age, sex, indication for surgery, operation, number and diameter of ports used, duration of surgery, intraoperative and postoperative complications, duration of hospitalization.